CLINICAL TRIAL: NCT02927418
Title: Strength Training for Injury Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS20030
Record Dates: First submitted 2016-10-05; First posted 2016-10-07 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2016-10

CONDITIONS: Wounds and Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength & Conditioning (Experimental): Supervised S & C program based on the Long Term Athlete Development Model. Participants will attend 2-3 sessions per week for about one hour each session for 4 months. The comprehensive program will include strength and power training as well as plyometrics, agility and flexibility exercises.
  Interventions: Behavioral: Strength & Conditioning
- Control (Active Comparator): Athletes in the control group will continue with their usual sports and activities but will not receive any type of training.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Strength & Conditioning
  Arms: Strength & Conditioning
Behavioral: Control
  Arms: Control

SUMMARY:
The purpose of this study is to explore the effects of a strength & conditioning (S & C) program on risk factors for injury (Y-balance and Functional Movement Screen scores), as well as parent reported injury occurrence in 12-16 year old male and female athletes. Forty girls and 40 boys aged 12-16 will be recruited; half will participate in supervised S & C sessions 2-3x/week while the other half will continue with their regular sports and activities. Risk factors for injury and performance indices (20 m sprint and multiple jump test) will be assessed before and after the 4 month study. Injury occurrence will be recorded via bi-weekly phone calls to the parent and athlete.

ELIGIBILITY:
Inclusion Criteria:

* Athletes between 12 and 16 years of age, actively participating in organized sport

Exclusion Criteria:

* Any condition or injury that will place the athlete at risk during testing or training

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-04-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Y-balance score | 4 months
  Using the Y Balance Test Kit (Functional Movement Systems, Inc., Chatham, Virginia), the athlete stands on one leg, hands on hips, while pushing a wooden block as far forward as possible with the opposite foot. The displacement of the block is recorded. The athlete is allowed 4 practice trials in each of the 3 test directions: anterior, posteromedial and posterolateral. Three test trials are then conducted for each leg in each direction, with short rest breaks between trials. The average reach distance for each leg for each direction will be normalized to leg length and used in analyses. This test has shown moderate to excellent reliability. Lower scores and asymmetries on the Y-balance test have been linked with an increased risk of injury.

SECONDARY OUTCOMES:
20 metre sprint | 4 months
  Athletes will perform 3 trials of a 20 metre sprint, with their time at 10 m and 20 m recorded. Timing will be done using a photo-electric timing system (SmartSpeed Pro, Fusion Sports, Chicago, USA). Each subject will wear a radio-frequency identification (RFID) bracelet assigned at the Open House sign-in; this device will allow timing for the sprint test. The fastest of the 3 trials will be used in analysis.
Multiple Jump test | 4 months
  Athletes will perform 3 different types of jumps. For each of the jumps the athlete stands on a Smart Jump Mat (SmartJump, Fusion Sports, Chicago, USA), and holds a dowel across the shoulders, behind the head. A static jump requires the athlete to crouch down for a jump, pause at the bottom, and then jump as high as possible. A countermovement jump requires the athletes to crouch down and immediately jump back up for maximum height. Three submaximal practice trials of each jump will be done, followed by 3 test trials. The goal is maximum vertical jump, measured by time in the air. Then a series of elastic jumps, maximizing height but minimizing time on the mat, will be done for 60 seconds. The athletes will have a short, submaximal practice trial first. The jump tests will allow for a description of the athletes' power qualities, which are important for sport performance.
Functional Movement Screen score | 4 months
  The FMS is a series of 7 tests including deep squat, hurdle step, in-line lunge, shoulder mobility, active straight leg raise, trunk stability push-up, and rotary stability tests. The intent of the test is to screen athletes for the ability to complete functional activities that underlie more complex athletic skills. A low score on the FMS has been related to increased injury risk.
Self-reported injury rates | 4 months
  Injury rates will be recorded during the study period by asking parents to contact the researcher when an injury occurs. A research assistant will also make bi-weekly phone calls to the parents/athletes in the study to ask about injury occurrence to ensure all injuries are noted. The type of injury (acute or overuse), involved body part, and treatment received will be documented as reported by the parent. No health identification numbers will be collected or healthcare practitioners contacted.

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Parsons, PhD, Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: No